CLINICAL TRIAL: NCT06044987
Title: The Effect of Concurrent Cystocele Repair on Transobturator Tape in Patients With Stress Urinary Incontinence - A Comparative Study
Brief Title: Effect of Cystocele Repair With Trans Obturator Tape VS. Trans Obturator Tape Alone on Stress Urinary Incontinence.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After discussing this study with the investigators, it was decided to consider it a retrospective study rather than a clinical trial. Since we could not delete this record, we chose the termination status instead.
Sponsor: Al-Mustafa University College (Other)
Collaborators: Al-Sadr Teaching Hospital (Other Government)
Responsible Party: Principal Investigator, Hayder Adnan Fawzi, Assistant Prof., Al-Mustafa University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-202301
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Stress Urinary Incontinence
Keywords: Urinary Incontinence, Stress; Cystocele; Trans Obturator Tape; Pelvic Organ Prolapse
MeSH Terms: conditions — Urinary Incontinence, Stress; Cystocele; Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (TOT alone) (Active Comparator): 49 Female Patients diagnosed with Stress urinary incontinence and cystocele and offered repair by Trans obturator tape procedure
  Interventions: Procedure: Trans Obturator Tape Procedure (TOT)
- Group II (TOT+ Cystocele Repair) (Experimental): 49 Female Patients diagnosed with Stress urinary incontinence and cystocele and offered repair by Trans obturator tape procedure concurrently with cystocele repair.
  Interventions: Procedure: Trans Obturator Tape Procedure (TOT); Procedure: Cystocele Repair

INTERVENTIONS:
Procedure: Trans Obturator Tape Procedure (TOT) — Done under Spinal anesthesia in the dorsal lithotomy position.
Procedure: Cystocele Repair — Done under Spinal anesthesia in the dorsal lithotomy position..
  Arms: Group II (TOT+ Cystocele Repair)

SUMMARY:
The goal of this interventional study is to compare the effect of Concurrent cystocele repair and trans obturator tape (TOT) and TOT alone in a sample of Iraqi Female participants with diagnosed stress urinary incontinence and cystocele. The main questions to answer are:

1-What are the effects of the tested Interventions on the outcomes measured by The Pelvic Organ Prolapse Quantification (POP-Q) System?

1. What are the effects of the tested Interventions on the degree of pelvic organ prolapse?
2. What are the effects of the tested Interventions on the frequency, severity, and effect of Stress urinary incontinence on the quality of life of the patients?
3. What are the effects of the tested Interventions on the impact of lower urinary tract symptoms on the quality of the patient's life?

Female Patients diagnosed with SUI indicated for intervention were divided into 2 groups

Group I: (n=49) offered TOT alone

Group II: (n=49) offered concurrent TOT and Cystocele Repair

Patients were then followed up and evaluated using The Pelvic Organ Prolapse Quantification (POP-Q) System, The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), and the King Health Questionnaire (KHQ). The efficacy of both procedures and their impact on SUI and quality of life was measured.

ELIGIBILITY:
Inclusion Criteria:

* Female patients.
* Pure stress and/or stress-predominant mixed urinary incontinence (MUI) associated with cystocele.
* Had not undergone a previous SUI surgery.
* BMI less than 35 kg/m2

Exclusion Criteria:

* Patients out of the age limit.
* Patients refused to participate in the study.
* Severe comorbid disease (heart failure HYHA class II and above, etc.).
* Patients with a previous surgical history of transvaginal mesh.
* Patients suffering detrusor overactivity.
* Patients diagnosed with the female genital system or urinary bladder Malignancies.
* Patients diagnosed with the presence of neurological disorders that caused voiding dysfunction.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Degree of Pelvic organ Prolapse (POP-Q) | At baseline, and at 9 months
  Assessed using the pelvic organ prolapse quantification system, in which it classified into:
  1. Stage 0: No prolapse is observed
  2. Stage 1: The most proximal portion of prolapse is greater than 1 cm above the level of the hymen
  3. Stage 2: The most proximal portion of prolapse is found between 1 cm higher than hymen and 1cm beneath hymen
  4. Stage 3: The most distal part of the prolapse extends more than 1cm beneath the hymen but no further than 2 cm
  5. Stage 4: vaginal eversion has taken place or eversion to with 2cm of TVL
Frequency, severity, and effect of urine incontinence on quality of life. | At baseline, and at 9 months
  Assessed using the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-SF). The score runs from "0 to 21", with higher values indicating more severe illness

SECONDARY OUTCOMES:
Impact of lower urinary tract symptoms including urinary incontinence on health-related quality of life. | At baseline, and after 9 months
  Assessed using the King Health Questionnaire (KHQ). It contains ten patient-rated domains. Each score value from 0% (best outcome) to 100% (worst outcome), except for Q10 from "0 to 30" with 30 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Hayder Adnan Fawzi, Ph.D, Study Chair — Al-Mustafa University College; Thaer Saleh Sabor Al-Omary, Ph.D, Principal Investigator — Al-Sadr Teaching Hospital
Locations (1):
- Al-Sadr Teaching Hospital, Amarah, Maysan Governorate, Iraq